CLINICAL TRIAL: NCT04787783
Title: Preanestes@s Phase 2. Evaluation of the Utility of a Web Based Application for Preoperative Care: Comparison of the Rate of Suboptimal Web-Based Assessments Versus the Outpatient Visit
Brief Title: Evaluation of the Utility of Preanestes@s, a Web Based Application for Preoperative Assessment
Acronym: Preanestes@s
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Preanestes@s. Phase2
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Mobile Applications; Internet-Based Intervention; Ambulatory Surgical Procedures; Preoperative Period
Keywords: Electronic Health Records; Patient Health Questionnaire; Health Impact Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web based assessment (Experimental): Participants will be leaded through preoperative period on a web based application. Participants will be addressed to either virtual or traditional face to face outpatient consultation on the basis of the information registered in the web based preoperative questionnaire that the application incorporates. Virtual assessment will be the performed by evaluating both the filled web based questionnaire together with participants´ electronic records. Face to face assessment will be performed in the traditional way by means of an interview with the participant together with the consultation of participant´s previous electronic records.
  Interventions: Other: Web based preoperative assessment
- Traditional face to face assessment (No Intervention): Participants will be leaded through preoperative period following traditional institutional standards of care.
  Face to face assessment will be performed in the traditional way by means of an interview with the participant together with the consultation of participant´s previous electronic records.

INTERVENTIONS:
Other: Web based preoperative assessment — Preoperative assessment conducted through a web based application
  Other Names: Preanestes@s
  Arms: Web based assessment

SUMMARY:
In this prospective two-arm study, the investigators will evaluate the incidence of suboptimal preoperative assessments when the participants are evaluated through a web based application (Preanestes@s) versus the traditional outpatient interview.

DETAILED DESCRIPTION:
Preanestes@s is a web based application conceived to lead patients through the preoperative period. The application includes a patient interface which offers general and individualized information on the perioperative process, with the possibility of generating a dynamic interaction between patients and medical staff. Patient interface incorporates a web based preoperative questionnaire that once fully completed automatically indicates which preoperative tests are necessary and addresses patients to a virtual (non face to face) consultation or to traditional outpatient assessment. Both virtual and outpatient assessment are performed by an anesthesiologist. The web based questionnaire automatically assigns patients an ASA (from the American Society of Anesthesia Physical Status Classification) grade; this being a determining variable, although not the only one, when directing patients to the virtual or face-to-face consultation.The questionnaire therefore serves both for collection of clinical information and as a patient classification tool as well.

Virtual assessment is performed by evaluating both the filled web based questionnaire together with patient´s electronic records. Face to face assessment is performed in the traditional way by means of a clinical interview together with the consultation of patient's previous electronic records.

The virtual assessment is reserved for participants without significant comorbidity, which would correspond to patients classified as grade ASA 1-2; this means without diseases or with diseases that do not significantly compromise the integrity of the patient: well-controlled hypertension, active smoking without major lung disease, non-morbid obesity, etc. Patients with significant comorbidity (grade ASA ≥ 3), are referred to a face-to-face consultation.

This study has been approved by the local Ethics Committee -Comité de Ética e Investigación de Huelva-and signed by its Secretary María Dolores Santos Rubio, date 18.12.2019, and corresponds to the Phase 2 of the study "Evaluation of the utility and quality of the clinical information obtained through Preanestes@s, a web based application for preoperative assessment. Comparison of the virtual preanesthetic visit and the outpatient face-to-face visit.". Phase 2 is independent of Phase 1, entitled "Evaluation of the Quality of Preoperative Information Obtained Through Preanestes@s, a Web Based Application: Paired Comparison of a Web Based Questionnaire, a Virtual Non Face to Face Assessment and Outpatient Visit", registered in Clinical Trials with number of reference NCT04259268. Primary completion of Phase 1 have been concluded with date February 19, 2021, and preliminary analysis of data is currently being conducted by investigators.

In this study, the objective of the investigators is to assess whether the use of a web based application for the preoperative assessment allows an adequate completion of the preoperative process when compared to traditional face to face outpatient interview. The quality of the information recorded by this web based application has been previously tested by the investigators showing promising results in terms of security and accuracy.

The investigators have designed a prospective two-arm study to compare the performance of the two modalities of preoperative assessment: web based versus face to face outpatient visit.

The investigators will base their evaluation of performance on previously published criteria: the Andalusian Regional Government Health Council defines a "suboptimal preoperative assessment" (SOPA) as one that potentially generates "inadequate preparation of the patient that may affect the expected results". Specific criteria defining SOPA are detailed in the Outcomes Measures section of the present document.

Allocation of participants to each study arm will be consecutive and based on daily distribution of the clinics: participants submitted to one of two surgeries of any of the following (Orthopedics, General Surgery, ENT) will be allocated to either web based preoperative assessment or traditional face to face outpatient visit. Written informed consent will be obtained of all participants prior to their recruitment.

Statistical analysis Data collection and subsequent analysis will be performed by the investigators team. Qualitative variables will be represented through the absolute and marginal frequencies. The investigators will analyze the incidence of SOPA in both groups, using Chi square to study the difference between the proportions in the case of normal distribution, or, failing that, the Mann-Whitney U. In the same way, the investigators will study the differences for each of the defining criteria of SOPA.

Sample Size Following the model of Kinley et al in the study comparing the quality of the pre-anesthesia record carried out by anesthesia trainees versus trained nurses, the investigators will use the variable "incomplete studies that could have affected perioperative management" for the calculation of the sample size. This variable would be equivalent to the variable SOPA in present work. Based on Kinley data, the investigators will use an incomplete study rate of 15%, a figure that coincides with the standard "inadequate assessment" in the Guide for the Perioperative Process published by the Andalusian Regional Government Health Council, which establishes a maximum "acceptable" rate of inadequate completion of the preoperative protocols in 15%. In this study of equivalence between the two formats, the investigators will assume equivalence if a maximum difference of 25% between both formats is observed, which represents a differential of 3.75% over the initial 15%. Thus, for a two-sided calculation and assuming an alpha error of 0.05 and a beta error of 0.2 (80% power), it would be necessary to include 1,127 participants per group.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing day surgery in our institution: Hospital Duques del Infantado, from Hospital Universitario Virgen del Rocío
* surgical specialities included: ENT, general surgery, orthopedics

Exclusion Criteria:

* Urgent procedures, patients without the ability to understand informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2254 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Suboptimal preoperative assessments (SOPA). | From the day of intervention up to 7 days after intervention
  Dichotomous (present/absent) composite variable comprising all possible causes of a predefined suboptimal result.
  Presence of any of the following:
  1. Lack of relevant information in the preoperative assessment that conducts to:
     * Inadequate conciliation of chronic medication
     * Inadequate preoperative fasting
     * Inadequate register of clinical or functional conditions that may cause delayed intervention the day of surgery (presence of uncontrolled chronic diseases, presence of impaired functional status undetected in the preoperative assessment, etc)
  2. Lack of complementary tests indicated according to preoperative protocol
  3. Presence of not indicated complementary tests according to preoperative protocol
  4. Lack of properly filled informed consent
  5. Cancellation of the intervention due to inadequate preoperative preparation (attributable to mismanagement of preoperative information-and analyzed by an expert´s committee )

CONTACTS AND LOCATIONS:
Overall Officials: Manuel de la Matta, MD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Hert S, Staender S, Fritsch G, Hinkelbein J, Afshari A, Bettelli G, Bock M, Chew MS, Coburn M, De Robertis E, Drinhaus H, Feldheiser A, Geldner G, Lahner D, Macas A, Neuhaus C, Rauch S, Santos-Ampuero MA, Solca M, Tanha N, Traskaite V, Wagner G, Wappler F. Pre-operative evaluation of adults undergoing elective noncardiac surgery: Updated guideline from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2018 Jun;35(6):407-465. doi: 10.1097/EJA.0000000000000817. PMID 29708905
- [Background] Pajuelo-Gallego A. Consejería de Salud, Junta de Andalucía. Bloque Quirúrgico: proceso de soporte. 2004. https://www.juntadeandalucia.es/organismos/saludyfamilias/areas/calidad-investigacion-conocimiento/gestion-conocimiento/paginas/pai-bloque-quirurgico.html
- [Background] Zaballos M, Lopez-Alvarez S, Argente P, Lopez A; Grupo de Trabajo de Pruebas Preoperatorias. Preoperative tests recommendations in adult patients for ambulatory surgery. Rev Esp Anestesiol Reanim. 2015 Jan;62(1):29-41. doi: 10.1016/j.redar.2014.07.007. Epub 2014 Aug 18. English, Spanish. PMID 25146773
- [Background] Blanco Vargas D, Faura Messa A, Izquierdo Tugas E, Santa-Olalla Bergua M, Noguera Sopena MM, Manoso Noriego M. [Online versus non-standard face to face preoperative assessment: cost effectiveness]. Rev Esp Anestesiol Reanim. 2012 Aug-Sep;59(7):350-6. doi: 10.1016/j.redar.2012.05.039. Epub 2012 Jul 10. Spanish. PMID 22784647
- [Background] Goodhart IM, Andrzejowski JC, Jones GL, Berthoud M, Dennis A, Mills GH, Radley SC. Patient-completed, preoperative web-based anaesthetic assessment questionnaire (electronic Personal Assessment Questionnaire PreOperative): Development and validation. Eur J Anaesthesiol. 2017 Apr;34(4):221-228. doi: 10.1097/EJA.0000000000000545. PMID 27798453
- [Background] National Guideline Centre (UK). Preoperative Tests (Update): Routine Preoperative Tests for Elective Surgery. London: National Institute for Health and Care Excellence (NICE); 2016 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK355755/ PMID 27077168
- [Background] Lozada MJ, Nguyen JT, Abouleish A, Prough D, Przkora R. Patient preference for the pre-anesthesia evaluation: Telephone versus in-office assessment. J Clin Anesth. 2016 Jun;31:145-8. doi: 10.1016/j.jclinane.2015.12.040. Epub 2016 Apr 15. PMID 27185698
- [Background] Kinley H, Czoski-Murray C, George S, McCabe C, Primrose J, Reilly C, Wood R, Nicolson P, Healy C, Read S, Norman J, Janke E, Alhameed H, Fernandes N, Thomas E. Effectiveness of appropriately trained nurses in preoperative assessment: randomised controlled equivalence/non-inferiority trial. BMJ. 2002 Dec 7;325(7376):1323. doi: 10.1136/bmj.325.7376.1323. PMID 12468478